CLINICAL TRIAL: NCT01334658
Title: Study of Endothelial Cell Density of Corneas Undergoing Phacoemulsification Surgery Using Balanced Salt Solution (BSS ®) Versus Glucose-bicarbonate-Ringer Lactate as Irrigating Solution: a Randomized Clinical Trial.
Brief Title: Study of Corneas Undergoing Balanced Salt Solution(BSS ®) Versus Glucose-bicarbonate-Ringer Lactate in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Estudos em Oftalmologia Clínica e Cirúrgica (Other)
Collaborators: CLIHON (Unknown)
Responsible Party: Hermelino Lopes de Oliveira Neto, GEOCC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100
Record Dates: First submitted 2011-04-08; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Cataract
Keywords: Corneal endothelium; Cataract surgery; Irrigation solutions intraocular; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balanced Salt Solution (BSS®) (Active Comparator): Subjects who received Balanced Salt Solution.
  Interventions: Procedure: Phacoemulsification cataract surgery; Drug: Balanced Salt Solution (BSS®)
- Glucose-bicarbonate-Ringer Lactate (GBRL) (Active Comparator): Subjects who received glucose-bicarbonate-Ringer Lactate.
  Interventions: Procedure: Phacoemulsification cataract surgery; Drug: Glucose-bicarbonate-Ringer Lactate (GBRL)

INTERVENTIONS:
Procedure: Phacoemulsification cataract surgery — A group received BSS ® (ALCON LABORATORIES, INC.) and another group received glucose-bicarbonate-Ringer Lactate (GBRL) [500 cc. Ringer Lactate (GLICOLABOR, Pharmaceutical LTD.) enriched with 1.5 ml of glucose in water (25%) and 08 ml of sodium bicarbonate (8.4%)] as a solution for irrigation during surgery.
  All surgeries were performed by single surgeon (HON), using the standard surgical technique quick-chop. Immediately before surgery, solutions for irrigation [BSS ® (ALCON LABORATORIES, INC..) and glucose-bicarbonate-Ringer Lactate (GBRL)] were brought to the operating table in a temperature of 22 degrees Celsius. The microcoaxial Phacoemulsification was performed under a phaco Legacy Series 20000 (ALCON LABORATORIES, INC..).
Drug: Glucose-bicarbonate-Ringer Lactate (GBRL) — A group received BSS ® (ALCON LABORATORIES, INC.) and another group received glucose-bicarbonate-Ringer Lactate (GBRL) [500 cc. Ringer Lactate (GLICOLABOR, Pharmaceutical LTD.) enriched with 1.5 ml of glucose in water (25%) and 08 ml of sodium bicarbonate (8.4%)] as a solution for irrigation during surgery.
  All surgeries were performed by single surgeon (HON), using the standard surgical technique quick-chop. Immediately before surgery, solutions for irrigation [BSS ® (ALCON LABORATORIES, INC..) and glucose-bicarbonate-Ringer Lactate (GBRL)] were brought to the operating table in a temperature of 22 degrees Celsius. The microcoaxial Phacoemulsification was performed under a phaco Legacy Series 20000 (ALCON LABORATORIES, INC..).
  Arms: Glucose-bicarbonate-Ringer Lactate (GBRL)
Drug: Balanced Salt Solution (BSS®) — A group received BSS ® (ALCON LABORATORIES, INC.) and another group received glucose-bicarbonate-Ringer Lactate (GBRL) [500 cc. Ringer Lactate (GLICOLABOR, Pharmaceutical LTD.) enriched with 1.5 ml of glucose in water (25%) and 08 ml of sodium bicarbonate (8.4%)] as a solution for irrigation during surgery.
  All surgeries were performed by single surgeon (HON), using the standard surgical technique quick-chop. Immediately before surgery, solutions for irrigation [BSS ® (ALCON LABORATORIES, INC..) and glucose-bicarbonate-Ringer Lactate (GBRL)] were brought to the operating table in a temperature of 22 degrees Celsius. The microcoaxial Phacoemulsification was performed under a phaco Legacy Series 20000 (ALCON LABORATORIES, INC..).
  Arms: Balanced Salt Solution (BSS®)

SUMMARY:
This is a study aimed at evaluating the effectiveness and impact of two intraocular irrigating solution (BSS ® versus glucose-bicarbonate-Ringer Lactate - GBRL) on the health of the cornea after cataract surgery by phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated senile cataract
* Visual acuity (VA) between 20/40 and 20/400
* Healthy corneas

Exclusion Criteria:

* Mental incapacity
* Patients with coexisting diseases of the cornea
* Presence of corneal opacity
* Uncontrolled glaucoma
* Uncontrolled diabetes mellitus
* Uveitis
* Cells or flare in the anterior chamber
* Prior intraocular surgery
* Patients using topical steroids or systemic
* Traumatic cataract, hereditary or toxic

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Increase in central corneal thickness (CCT) | Two days after surgery.
Increase in central corneal thickness (CCT) | Thirty days after surgery.
Increase in central corneal thickness (CCT) | Ninety days after surgery.
Decrease in the percentage of endothelial cell density (ECD) | Two days after surgery.
Decrease in the percentage of endothelial cell density (ECD) | Thirty days after surgery.
Decrease in the percentage of endothelial cell density (ECD) | Ninety days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hermelino L Oliveira Neto, Study Director — CLIHON; Israel C Marques Neto, Principal Investigator — State University of Feira de Santana (UEFS); Brunno B Barros, Principal Investigator — State University of Feira de Santana (UEFS)